CLINICAL TRIAL: NCT00717509
Title: Cross-Sectional Study of the Association Between Multiple Genetic Polymorphisms and the Metabolic Side Effects in Patients With Schizophrenia Taking Clozapine More Than 1 Year
Brief Title: Association of Multiple Genetic Polymorphisms With Clozapine-Associated Metabolic Change in Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National Hospital (Other Government)
Responsible Party: Shi Hyun Kang, Seoul National Hospital
Other Study IDs: snh003
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Schizophrenia; Metabolic Syndrome; Genetic Polymorphism
Keywords: schizophrenia; metabolic side effect; clozapine; genetic polymorphism
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- clozapine group: * chronic schizophrenia
  * have been taking clozapine at leaset one year
  * without diabetes, pulmonary tuberculosis

SUMMARY:
We are going to investigate the association of multiple genetic polymorphisms with the metabolic side effects in patients with schizophrenia taking clozapine.

DETAILED DESCRIPTION:
The use of antipsychotics, especially clozapine and olanzapine is associated with metabolic side effects, which put patients with schizophrenia at risk for cardiovascular morbidity or diabetes.

The prevalence of the metabolic syndrome was 53.8% of patients who taking clozapine. The high interindividual variability in antipsychotic-induced metabolic abnormalities suggests that genetic makeup is a possible determinant.

The genotypes of the multiple gene such as HTR2C, LEP, adrenergic receptor,PPAR,GNB3 are suggested to have associations with the metabolic side effects (weight,glucose,lipid,BP,metabolic syndrome) in patients using antipsychotics.

We are going to investigate whether those multiple genetic polymorphisms are associated with the metabolic side effects in patients taking clozapine.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* who can understand and sign the informed consent

Exclusion Criteria:

* who refuse to participate this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with schizophrenia taking clozapine more than 1 year
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-01 (Actual); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
The associations between multiplegenetic polymorphisms (HTR2C,leptin,adrenergic receptor,PPAR,GNB3) and the metabolic side effects (weight,glucose,lipid,BP,metabolic syndrome) | more than 1 year after starting clozapine

CONTACTS AND LOCATIONS:
Overall Officials: Shi Hyun Kang, M.D., Study Director — Seoul National Hospital
Locations (1):
- Seoul National Hospital, Seoul, South Korea